CLINICAL TRIAL: NCT00646568
Title: hCG Stimulating Test of the Thecal Cells to Evaluate the Ovarian Reserve
Brief Title: Human Chorionic Gonadotropin (hCG) Test: A Novel Method to Evaluate the Ovarian Reserve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Arik Tzukert, Hadassah Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: hcgstimtest-HMO-CTIL
Record Dates: First submitted 2008-03-17; First posted 2008-03-28 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Infertility
Keywords: IVF; ovarian reserve; androgens; thecal cells; Fertility Agents, Female
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

INTERVENTIONS:
Drug: s.c. human chorionic gonadotropin (Pregnyl) — S.C. Pregnyl 10000 IU once

SUMMARY:
In an era of delayed fertility plans, there is an increasing need for a reliable method to predict ovarian reserve and responsiveness. The current tests include serum FSH, Inhibin B, Mullerian inhibiting factor (MIF) and ultrasonographic measures such as ovarian volume and number of antral follicles are non-specific and with questionable reliability. The biochemical tests represent the function of production of androgens, as a predictor of ovarian reserve, has not been tested yet.

Working hypothesis and aims: testing the prognostic capability of hCG stimulating test of theca cells for estimating the ovarian reserve, and by that to calculate better the chance for IVF cycle success

DETAILED DESCRIPTION:
20 women >40 years old and 20 women <35 years old, attended to our IVF unit were included in the study. Another 20 other young women (<35 years) with poor response in previous IVF cycles will be participate. All participants received a single hCG 10000 IU injection on cycle day 2-4. Hormone levels of LH, FSH, E2, P, Testosterone, Androstendione and 17-OHP were taken prior to the injection and on days 1, 3 and 7 afterwards. hCG induced hormone levels will be compared with IVF results

ELIGIBILITY:
Inclusion Criteria:

* All women on IVF cycle

Exclusion Criteria:

* Any allergy to injection of human chorionic gonadotropin before

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
androgens levels after stimulation in relation to the ovarian reserve | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Assaf Ben-Meir, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical center, Jerusalem, Israel